CLINICAL TRIAL: NCT02227485
Title: Evaluation of the Effects of an Iranian Traditional Mouth Rinse Punica Granatum Pleniflora (Golnaar) in Treatment of Gingivitis in Patients With Diabetes Mellitus
Brief Title: Iranian Traditional Mouth Rinse Punica Granatum Pleniflora (Golnaar) in Treatment of Gingivitis in Diabetic Patients
Acronym: Golnaar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of Internal Medicine & Endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT93747064
Record Dates: First submitted 2014-08-22; First posted 2014-08-28 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Gingivitis
Keywords: Gingivitis; Diabetes mellitus; Medicine, Traditional; Herbal medicine; Punica granatum
MeSH Terms: conditions — Gingivitis; Diabetes Mellitus | interventions — Mouthwashes; Chlorhexidine; Control Groups; Tooth Bleaching

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine (0.2%) (Active Comparator): Chlorhexidine (0.2%) mouth rinse, 10 ml for 2 minutes every night for 2 weeks and tooth bleaching (one time) after using mouth rinse.
  Interventions: Drug: Chlorhexidine (0.2%); Procedure: Tooth bleaching
- Punica granatum Pleniflora mouth rinse (Experimental): Punica granatum Pleniflora (Golnaar) mouth rinse, 10 ml for 2 minutes every night for 2 weeks and tooth bleaching (one time) after using mouth rinse.
  Interventions: Drug: Punica granatum Pleniflora (Golnaar) mouth rinse; Procedure: Tooth bleaching

INTERVENTIONS:
Drug: Punica granatum Pleniflora (Golnaar) mouth rinse — All the patient in intervention group use 10 ml of "Golnaar" mouth rinse for 2 minutes every night for 2 weeks.
  Other Names: Intervention group
  Arms: Punica granatum Pleniflora mouth rinse
Drug: Chlorhexidine (0.2%) — All the patient in control group use 10 ml of chlorhexidine (0.2%) for 2 minutes every night for 2 weeks.
  Other Names: Control group
  Arms: Chlorhexidine (0.2%)
Procedure: Tooth bleaching — Tooth bleaching for both groups one time after using mouth rinses.
  Other Names: Bleaching

SUMMARY:
This is a triple-blinded randomized clinical trial to evaluate the effect of an Iranian traditional mouth rinse (Punica granatum Pleniflora or "Golnaar" mouthrinse) on treatment of diabetic gingivitis and compare it with chlorhexidine (0.2%).

DETAILED DESCRIPTION:
Among diabetic patients who refer to Motahhari clinic of Shiraz University of Medical Sciences 80 volunteers who have gingivitis and aged between 20 to 65 years old and fulfill other inclusion criteria, are randomly assigned to intervention or control groups. All of the patients will undergo a training panel about mouth hygiene and receive a pack of a toothbrush, a toothpaste, a dental floss and a mouth rinse. They are asked to return after 2 weeks for the second evaluation and taking tooth bleaching. The demographic and general information of all participants are taken and the primary outputs (plaque index and bleeding on probe) are measured at the beginning, after 2 weeks and after 4 weeks. All the examinations are done by one trained person and patients, practitioner and statistical analyser are blind to the interventions.

ELIGIBILITY:
Inclusion Criteria:

* To have gingivitis
* Controlled diabetes mellitus [FBS<130mg/dl & Glycosilated hemoglobin (A1C)<7%]
* Presence of gingivitis
* Having at least 20 teeth
* No history of hypersensitivity reaction
* Age between 20 to 65 years
* Agreement to participate in the study

Exclusion Criteria:

* History of hypersensitivity reaction
* Smoking
* Systemic diseases (Kidney, liver or rheumatologic diseases)
* To have a pocket depth of more than 5
* Consumption of antibiotics, corticosteroids or nonsteroidal anti-inflammatory drugs in the past 3 months and during the study period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mesbah Shams, MD, Study Chair — Research Center for Traditional Medicine & History of Medicine - Shiraz University of Medical Sciences; Mohammad Mahdi Fani, Dentist, Principal Investigator — Research Center for Traditional Medicine & History of Medicine-Shiraz University of Medical Sciences; Massih Seddigh-Rahimabadi, MD, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Motahhari clinic of Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Yes
All the records have been collected and archived, and can be reused if is necessary.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for Chlorhexidine group started on 11/05/2014 and ended on 07/11/2014. For Golnaar group the starting and ending dates were; 01/05/2014 and 09/11/2014.
Period: First Follow-up
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Started | 40 | 40
Completed | 36 (At the first follow-up we lost 4 patients.) | 38 (After 2 weeks, 2 patients had withdrew the study.)
Not Completed | 4 | 2
Period: Second Follow-up
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Started | 36 | 38
Completed | 34 (At the second follow-up we lost 2 patients.) | 36 (At the second follow-up we lost 2 patients.)
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Chlorhexidine (0.2%): Chlorhexidine (0.2%) mouth rinse, 10 ml for 2 minutes every night for 2 weeks and tooth bleaching (one time) after using mouth rinse.
  Chlorhexidine (0.2%): All the patients in control group use 10 ml of chlorhexidine (0.2%) for 2 minutes every night for 2 weeks.
  Tooth bleaching: Tooth bleaching for both groups one time after using mouth rinses.
- Punica Granatum Pleniflora Mouth Rinse: Punica granatum Pleniflora (Golnaar) mouth rinse, 10 ml for 2 minutes every night for 2 weeks and tooth bleaching (one time) after using mouth rinse.
  Punica granatum Pleniflora (Golnaar) mouth rinse: All the patients in intervention group use 10 ml of "Golnaar" mouth rinse for 2 minutes every night for 2 weeks.
  Tooth bleaching: Tooth bleaching for both groups one time after using mouth rinses.
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (6.5) | 50.35 (6.9) | 51.33 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 40 | 40 | 80
Height [Mean (Standard Deviation); unit: cm] — The height of patients in centimeter (cm)
  cm | 163.9 (9.6) | 164.1 (10.0) | 164 (9.7)
Weight [Mean (Standard Deviation); unit: kg] | 75.1 (13.5) | 75.6 (13.8) | 75.4 (13.6)
Disease duration [Mean (Standard Deviation); unit: years] | 10.3 (6.2) | 9.7 (6.3) | 10 (6.2)
Teeth number [Mean (Standard Deviation); unit: teeth] | 24.7 (3.3) | 25.0 (3.6) | 24.9 (3.4)
BP [Mean (Standard Deviation); unit: mm Hg] — The maximum arterial blood pressure
  mm Hg | 12.3 (1) | 12.5 (1.2) | 12.4 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index
Description: 0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth, which cannot be seen with the naked eye. But only by using disclosing solution or by using probe.
  2. Moderate accumulation of deposits within the gingival pocket, on the gingival margin and/ or adjacent tooth surface, which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Time Frame: At the beginning, after 2 weeks and after 4 weeks
Population: The number of analysed cases for the base line section are 40 and for other sections (after 2 weeks and 4 weeks) are 34 for Chlorhexidine group and 36 for Punica granatum group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Chlorhexidine (0.2%): Chlorhexidine (0.2%) mouth rinse, 10 ml for 2 minutes every night for 2 weeks and tooth bleaching (one time) after using mouth rinse.
  Chlorhexidine (0.2%): All the patient in control group use 10 ml of chlorhexidine (2%) for 2 minutes every night for 2 weeks.
  Tooth bleaching: Tooth bleaching for both groups one time after using mouth rinses.
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Number analyzed (Participants) | 40 | 40
units on a scale
  At base line | 2.3 (0.9) | 2.5 (0.6)
  After 2 weeks | 1.9 (1) | 2 (0.7)
  After 4 weeks | 0.2 (0.2) | 0.2 (0.1)

2. Primary Outcome: Bleeding Index
Description: presence of bleeding of the gum when probing it: 0= No bleeding
  1= Bleeding occurs within 10 seconds after gentle probing of the orifice of the gingival crevice
Time Frame: At the beginning, after 2 weeks and after 4 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Number analyzed (Participants) | 40 | 40
units on a scale
  At base line | 0.133 (0.097) | 0.148 (0.123)
  After 2 weeks | 0.039 (0.057) | 0.034 (0.056)
  After 4 weeks | 0.01 (0.034) | 0.016 (0.03)

3. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Up to 2 weeks
Measure: Number; unit: participants
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Number analyzed (Participants) | 36 | 38
participants
  No adverse event | 15 | 22
  Had some adverse event | 21 | 16

4. Secondary Outcome: Satisfaction of Patients
Description: We use a Visual Analogue Scale (VAS) to evaluate the patients' satisfaction and their tolerance.
  This "VAS" ranged from 1 (not satisfied at all) to 5 (fully satisfied) was used:
  1. Not satisfied at all
  2. Not satisfied adequately
  3. Not good-Not bad (So So)
  4. Mostly Satisfied
  5. Fully satisfied
Time Frame: Up to 2 week
Measure: Number; unit: participants
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Number analyzed (Participants) | 36 | 38
participants
  Satisfied | 32 | 36
  Unsatisfied | 1 | 0
  So-So | 3 | 2

5. Primary Outcome: Pocket Depth
Description: It is the depth of the dental sulcus which detected by measuring the depth of sulcular insertion of the probe at six sites; mesiofacial, midfacial, distofacial, mesiolingual, midlingual and distolingual of all teeth divided by the teeth number. the measurement unit is millimeter (mm).
Time Frame: At the beginning, after 2 weeks and after 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Number analyzed (Participants) | 40 | 40
mm
  At base line | 1.3 (0.8) | 1.6 (1.1)
  After 2 weeks | 0.9 (0.7) | 0.8 (0.8)
  After 4 weeks | 0.6 (0.6) | 0.6 (0.7)

6. Primary Outcome: Modified Gingival Index
Description: 0= Absence of inflammation
  1. Mild inflammation or with slight changes in color and texture but not in all portions of gingival marginal or papillary
  2. Mild inflammation, such as the preceding criteria, in all portions of gingival marginal or papillary
  3. moderate, bright surface inflammation, erythema, edema and/or hypertrophy of gingival marginal or papillary
  4. severe inflammation: erythema, edema and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion or ulceration
Time Frame: At the beginning, after 2 weeks and after 4 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Number analyzed (Participants) | 40 | 40
units on a scale
  At base line | 1.3 (1) | 1.3 (0.9)
  After 2 weeks | 0.4 (0.6) | 0.2 (0.4)
  After 4 weeks | 0.1 (0.3) | 0 (0.1)

ADVERSE EVENTS:
Time Frame: During the study and up to 1 month after finishing mouth rinses.
Arm/Group | Chlorhexidine (0.2%) | Punica Granatum Pleniflora Mouth Rinse
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 21/36 | 16/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorhexidine (0.2%) (N=36) | Punica Granatum Pleniflora Mouth Rinse (N=38)
Unpleasant taste (Surgical and medical procedures) | 14 (14) | 15 (15)
Other side effects (Surgical and medical procedures) | 4 (4) | 0 (0)
Discolored (Surgical and medical procedures) | 3 (3) | 0 (0)
Bad Odor (Surgical and medical procedures) | 0 (0) | 1 (1) — Bad odor of the mouth wash

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes